CLINICAL TRIAL: NCT04969796
Title: Supporting Caregivers of Veterans With TBI and Mixed Dementia: The REACH Hope Behavioral Intervention
Brief Title: REACH Hope Intervention for Dementia and TBI Caregivers
Acronym: REACH Hope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Memphis VA Medical Center (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other); University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZ190094
Record Dates: First submitted 2021-07-01; First posted 2021-07-21 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Dementia, Mixed; Dementia of Alzheimer Type; TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Mixed Dementias; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: The study is a wait list control design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH Hope (Experimental): Participants receive the REACH behavioral intervention coupled with the Department of Defense Hope Box app.
  Interventions: Other: REACH Hope
- Wait list control (Active Comparator): Participants receive the REACH behavioral intervention coupled with the Department of Defense Hope Box app.
  Interventions: Other: REACH Hope

INTERVENTIONS:
Other: REACH Hope — REACH VA (Resources for Enhancing All Caregivers Health in Department of Veterans Affairs) and the DoD's Virtual Hope Box. For REACH Hope, as the caregiver and interventionist work on strategies one-on-one, these will be integrated into the Hope Box for the caregiver to use between and after sessions.

SUMMARY:
This three-year randomized clinical trial will evaluate a behavioral intervention for caregivers of Veterans with traumatic brain injury (TBI) and Alzheimer's dementia or mixed Dementia (AD/MD) to reduce caregiver depression, anxiety and burden, and improve veterans' health management. The study will combine and deliver two award-winning behavioral interventions - REACH VA (Resources for Enhancing All Caregivers Health in Department of Veterans Affairs) and the DoD's Virtual Hope Box, which we call REACH Hope. Both REACH and Hope Box have evidence of effectiveness individually but have not been delivered together for caregivers supporting veterans with complex neurodegenerative diagnoses and health conditions. Our primary hypothesis is that REACH Hope will improve caregivers' quality of life as measured by reduced burden.

ELIGIBILITY:
Inclusion Criteria:

* primary caregiver for person with diagnosis of TBI and subsequent dementia
* at least one activity of daily living limitation or 2 or more instrumental activity of daily living limitation
* provide 4 or more hours of care per day for at least 6 months
* endorse a score of at least high burden (>8) on the Zarit Burden Inventory-4

Exclusion Criteria:

* no mobile telephone or electronic device that can accept the Hope Box application
* current diagnosis of schizophrenia or other major mental illness
* auditory impairment that would make telephone use difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-14 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Burden at three months | three months
  Measured by the Zarit Burden Inventory- 12
Change from baseline Burden at six months | six months
  Measured by the Zarit Burden Inventory- 12

SECONDARY OUTCOMES:
Change from baseline Depression at three months | Three months
  As measured with the Patient Health Questionnaire-9
Change from baseline Depression at six months | Six months
  As measured with the Patient Health Questionnaire-9
Change from baseline Anxiety at three months | Three months
  As measured with the General Anxiety Disorders-7
Change from baseline Anxiety at six months | six months
  As measured with the General Anxiety Disorders-7
Change from baseline Caregiving self-efficacy at three months | three months
  As measured with the Caregiving Self-Efficacy scale
Change from baseline Caregiving self-efficacy at six months | six months
  As measured with the Caregiving Self-Efficacy scale

CONTACTS AND LOCATIONS:
Overall Officials: Linda O Nichols, PhD, Principal Investigator — US Department of Veterans Affairs; Paul Perrin, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Caregiver Center, VA Medical Center, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Nichols LO, Martindale-Adams J, Seel RT, Zuber JK, Perera R, Perrin PB. Reducing burden and anxiety for caregivers of veterans with traumatic brain injury and dementia: Randomized controlled trial of the resources for enhancing all caregivers' health-Hope intervention. Rehabil Psychol. 2025 Jul 31:10.1037/rep0000632. doi: 10.1037/rep0000632. Online ahead of print. PMID 40742769